CLINICAL TRIAL: NCT02159027
Title: Maraviroc and NeuroAIDS Pathogenesis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: ViiV Healthcare (Industry); University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H024
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: AIDS Dementia Complex
Keywords: Human Immunodeficiency Virus; AIDS Dementia Complex
MeSH Terms: conditions — AIDS Dementia Complex; Acquired Immunodeficiency Syndrome | interventions — Maraviroc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): placebo identical in appearance to maraviroc 150 and 300 mg tablets will be added to each subjects antiretroviral regimen at doses as recommended by the package insert
  Interventions: Drug: Placebo
- maraviroc (Experimental): Maraviroc Tablets are available as 150 mg and 300 mg tablets. Each subject will add maraviroc to their current antiretroviral regimen with dosage based on recommendations as per maraviroc package insert
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — Maraviroc administered twice daily, dosage based on concomitant medication being taken.
  Other Names: Selzentry
  Arms: maraviroc
Drug: Placebo — Maraviroc placebo administered twice daily, dosage based on concomitant medication being taken.
  Arms: placebo

SUMMARY:
Maraviroc is an antiretroviral medication that may help in improving mental function in HIV infected patients with mental problems by decreasing inflammatory tendencies. We will test this in a clinical trial of 42 HIV infected individuals with some mild to moderate mental problems who are already on HIV medications and doing well. We will add Maraviroc or a sugar pill to their HIV medications and see if mental function improves over 48 weeks. This study will be conducted at 2 sites in Hawaii and Puerto Rico.

DETAILED DESCRIPTION:
We hypothesize that maraviroc (MVC) will lead to improved cognition as assessed by improvement in neuropsychological (NP) performance. We hypothesize that MVC therapy leads to (1) decrease in HIV infection of monocytes (MO), particularly of CD16-expressing MO and (2) phenotypic and functional secretory changes suggestive of decrease in MO immune activation, and that these changes will lead to less HIV infected activated MO trafficking to the CNS, less CNS inflammation and neuronal damage, and ultimately improved cognition. We will test this in a 48 week trial in 42 HIV infected individuals on suppressive antiretroviral therapy (ART) with mild to moderate cognitive dysfunction. These individuals will be randomized to intensify their ART in double-blind fashion to MVC vs placebo. The primary endpoint will be change in NPZglobal. Magnetic resonance spectroscopy (MRS)/magnetic resonance spectroscopic imaging (MRSI) will be conducted to assess potential alterations in inflammatory and neuronal brain chemicals.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of HIV-1 infection by an FDA approved test at any time prior to study entry.
* Receipt of ARV medication uninterrupted for > 1 year leading up to the screening period; brief interruptions for toxicity purposes will be evaluated on a case by case basis and may be allowed
* Screening plasma HIV RNA < 50 copies/ml within 3 months of entry
* Willingness for both males and females of childbearing potential to utilize 2 effective contraception methods (2 separate forms, one of which must be an effective barrier method), be non-heterosexually active or have a an exclusive vasectomized partner from screening throughout the duration of the study treatment and for 30 days following the last dose of study drugs.
* Age between 18 to 70 years.
* Ability and willingness to provide written informed consent Mild to moderate cognitive impairment with global neuropsychological (NP) test (NPZglobal) score of < -0.5 OR a neurocognitive abnormality (< -0.5) in at least one cognitive domain known to be typically affected by HIV

Exclusion Criteria:

* Currently receiving or having used a CCR5 antagonist as part of an antiretroviral regimen within 6 months of study entry
* Plasma HIV RNA > 100 copies/ml at any time within 6 months of study entry
* History of HIV-2
* Diagnosis of cirrhosis
* Active or inadequately treated tuberculosis (TB) infection, or inadequate treatment for a positive purified protein derivative (PPD) test. Adequate treatment is defined as meeting the current recommendations of the Centers of Disease Control and Prevention (CDC), National Institutes of Health (NIH) and the HIV Medicine Association of the Infectious Diseases Society of America (IDSA) guidelines33 or other CDC recommendations if the patient was treated before the current recommendations or before coinfection with HIV.
* Uncontrolled seizure disorder
* Current malignancy or history of past malignancies excluding basal cell CA and Kaposi's sarcoma restricted to the skin, unless subject considered cured.
* Any immunomodulator, HIV vaccine, any other vaccine, or investigational therapy within 30 days of study entry.
* Requirement for acute therapy for any AIDS-defining illness or other serious medical illnesses (in the opinion of the site investigator) within 14 days prior to entry.
* Chronic illnesses including hematologic, pulmonary, and autoimmune diseases and endocrinopathies, except for stable controlled diabetes or cardiovascular disease in the view of the investigator and stable testosterone or thyroid medication use
* Known hypersensitivity to MVC or its excipients
* Anticipated need for specific prescription medications. Unwillingness to stop from eating grapefruit or using St. John's wort.
* Chronic use of over-the-counter (OTC) medications unless approved by Study Investigator
* Hemoglobin < 9.0; Absolute neutrophil count < 500/μL; Platelet count < 40,000/μL; AST (SGOT) and ALT (SGPT) > 5x ULN; Lipase > 2.0 x ULN
* Estimated creatinine clearance < 30 cc/min using Cockcroft and Gault method
* Abnormal EKG unless determined by the Investigator to be not clinically significant.
* Presence of any condition that would interfere with the absorption, distribution, metabolism, or excretion of the drug
* Current illicit substance or alcohol use or abuse which, in the judgment of the Investigator, will interfere with the patient's ability to comply with the protocol requirements
* Pregnancy or breast-feeding, intent to become pregnant during the study
* Patients, who, in the opinion of the Investigator, are unable to comply with the dosing schedule and protocol evaluation or for whom the study may not be advisable
* Any factor that precludes MRI scan including presence of metal or exposure to metal work (e.g. metal grinder/worker) and claustrophobia
* Any CNS pathology which, in the judgment of the investigator, will interfere with the ability to assess study change in MRSI
* Learning disability, history of head injury with prolonged loss of consciousness or cognitive sequelae, history of opportunistic infection of the brain or other non-HIV etiologies that, in the judgment of the investigator, can explain the subjects's mild to moderate cognitive performance.
* Serum B12 or folate below the lower limits of normal
* Abnormal TSH, except when free T4 is within normal limits
* History of untreated or inadequately treated positive RPR

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Change in Neuropsychological Performance | 48 weeks
  Change in global neuro-psychological Z scores and change in various neuro-psychological Z subdomains will be assessed

SECONDARY OUTCOMES:
Changes in monocyte subsets and function | 48 weeks
  Change in monocyte subsets based on CD14 and CD16 expression by flow cytometry; Change in inflammatory and neurotoxic mediators (sCD14, TNFalpha, sCD163 and neopterin
Change in HIV DNA content within MO subsets | 48 weeks
  Change in HIV DNA content specifically within each MO subsets
Change in brain metabolites by magnetic resonance spectroscopy | 48 weeks
  Change in neuronal and inflammatory brain metabolites globally within brain and in select brain regions

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia M. Shikuma, M.D., Principal Investigator — University of Hawaii
Locations (2):
- Clint Spencer Clinic, Hawaii Center for AIDS, University of Hawaii, Honolulu, Hawaii, United States
- Puerto Rico Clinical and Translational Research Consortium, San Juan, Puerto Rico

REFERENCES:
- [Result] Ndhlovu LC, Umaki T, Chew GM, Chow DC, Agsalda M, Kallianpur KJ, Paul R, Zhang G, Ho E, Hanks N, Nakamoto B, Shiramizu BT, Shikuma CM. Treatment intensification with maraviroc (CCR5 antagonist) leads to declines in CD16-expressing monocytes in cART-suppressed chronic HIV-infected subjects and is associated with improvements in neurocognitive test performance: implications for HIV-associated neurocognitive disease (HAND). J Neurovirol. 2014 Dec;20(6):571-82. doi: 10.1007/s13365-014-0279-x. Epub 2014 Sep 17. PMID 25227930